CLINICAL TRIAL: NCT05395091
Title: A Randomized, Double-Blind, Parallel Design, Repeat Dose, 2-arm, Multicenter Study Comparing the Efficacy, Safety, Immunogenicity, and Pharmacokinetic Profiles of AVT03 and US-Prolia® in Postmenopausal Women With Osteoporosis, ALVOBOND
Brief Title: Multicenter Study in Postmenopausal Women With Osteoporosis, ALVOBOND
Acronym: ALVOBOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alvotech Swiss AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVT03-GL-C01
Record Dates: First submitted 2022-05-24; First posted 2022-05-27 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Postmenopausal Osteoporosis, Denosumab, Alvotech
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- AVT03 (Experimental): AVT03 is the proposed biosimilar for Prolia.
  Interventions: Biological: AVT03
- Prolia (Active Comparator)
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: AVT03 — AVT03 (denosumab) is a recombinant fully human IgG2 monoclonal antibody to RANKL to be administered as a subcutaneous injection. Subjects in this arm received AVT03 60mg administered s.c. on Day 1 and at Month 6. At Month 12, subjects in the AVT03 arm received a third dose of AVT03 60 mg.
  Arms: AVT03
Biological: Denosumab — Prolia (denosumab) is a recombinant fully human IgG2 monoclonal antibody to RANKL developed to be administered as a subcutaneous injection.
  Subjects in this arm received 60mg of commercially available US-Prolia, administered s.c on Day 1 and at Month 6. At Month 12, subjects in the Prolia treatment group were re-randomized in a 1:1 ratio to receive either:
  * AVT03 60 mg administered s.c. on Day365.
  * Prolia 60 mg administered s.c. on Day365.
  Other Names: Prolia
  Arms: Prolia

SUMMARY:
This is a randomized, double-blind, parallel design, repeat dose, 2 arm, multicenter study comparing the efficacy, safety, immunogenicity, pharmacodynamic (PD) and pharmacokinetic (PK) profiles of AVT03 and US-Prolia in postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
After the screening activities, eligible subjects were randomized to receive either AVT03 60 mg or Prolia® 60 mg, administered as a subcutaneous (s.c.) injection on Day 1 and at Month 6. At Month 12, subjects in AVT03 treatment group will received a third dose of AVT03 60 mg administered s.c. while subjects in Prolia® treatment group will were be re-randomized 1:1 to receive either Prolia 60 mg or AVT03 60 mg administered as a subcutaneous injection.

Afterwards, the subjects will be followed until the End of Study (EoS) Visit.

ELIGIBILITY:
1. Postmenopausal women with osteoporosis willing to sign an informed consent form (ICF)and able to undergo protocol related procedures.
2. A baseline dual-energy x-ray absorptiometry (DXA) scan with a T score ≤-2.5 and

   * 4.0 at the LS (L1 to L4)and/or, total hip, and/or femoral neck.
3. Age: ≥50 years.
4. Female subject is postmenopausal according to 1 of the following criteria:

   1. Spontaneous amenorrhea for ≥12 consecutive months
   2. Biochemical criteria of menopause, follicle-stimulating hormone, >40 IU/L except surgically sterile
   3. Having had bilateral oophorectomy ≥6 weeks prior to Screening
5. Willing to receive calcium plus vitamin D supplements.
6. At least 2 consecutive evaluable lumbar vertebrae and at least 1 evaluable hip.

Exclusion Criteria

1. Evidence of clinically relevant pathology, especially prior diagnosis of bone disease, or any uncontrolled condition that will affect bone metabolism
2. History and/or presence of 1 severe or more than 1 moderate vertebral fractures confirmed by x-ray.
3. History of hip fracture
4. Presence of active healing fractures
5. Osteonecrosis of the jaw (ONJ) or risk factors for ONJ such as invasive dental procedures
6. Evidence of hypo/hypercalcemia at Screening
7. Known vitamin D deficiency
8. Known intolerance to calcium and vitamin D supplement.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felicitas Bullo, Study Director — Alvotech Swiss AG
Locations (34):
- Bulgaria (3):
  - Investigational Site 3501, Plovdiv
  - Investigational Site 3503, Plovdiv
  - Investigational Site 3502, Stara Zagora
- Czechia (2):
  - Investigational Site 4201, Prague
  - Investigational Site 4202, Uherské Hradiště
- Georgia (6):
  - Investigational Site 9901, Tbilisi
  - Investigational Site 9902, Tbilisi
  - Investigational Site 9903, Tbilisi
  - Investigational Site 9904, Tbilisi
  - Investigational Site 9905, Tbilisi
  - Investigational Site 9906, Tbilisi
- Poland (11):
  - Investigational Site 4803, Bialystok
  - Investigational Site 4804, Bialystok
  - Investigational Site 4802, Krakow
  - Investigational Site 4807, Krakow
  - Investigational Site 4806, Lodz
  - Investigational Site 4811, Lublin
  - Investigational Site 4812, Poznan
  - Investigational Site 4801, Skierniewice
  - Investigational Site 4805, Świdnik
  - Investigational Site 4809, Warsaw
  - Investigational Site 4810, Zamość
- South Africa (12):
  - Investigational Site 2705, Bloemfontein
  - Investigational Site 2714, Cape Town
  - Investigational Site 2707, Centurion
  - Investigational Site 2708, Centurion
  - Investigational Site 2710, Groenkloof
  - Investigational Site 2712, Johannesburg
  - Investigational Site 2702, KwaDukuza
  - Investigational Site 2711, Parow
  - Investigational Site 2701, Port Elizabeth
  - Investigational Site 2706, Pretoria
  - Investigational Site 2713, Pretoria
  - Investigational Site 2703, Worcester

REFERENCES:
- [Derived] Lortkipanidze M, de Villiers T, Kania G, Bullo F, Jaskiewicz L, Stamatakos S, Rai M, Haliduola H, Otto H, Sattar A, Leutz S, Berti F. A randomized, double blind, parallel design, repeat dose, 2-arm, multicenter study comparing the efficacy, safety, immunogenicity, and pharmacokinetic profiles of a denosumab biosimilar, AVT03, in postmenopausal women with osteoporosis. Expert Opin Biol Ther. 2025 Aug;25(8):899-912. doi: 10.1080/14712598.2025.2538609. Epub 2025 Jul 28. PMID 40698538

RESULTS

PARTICIPANT FLOW:
Groups:
- AVT03: AVT03 is a proposed biosimilar for Prolia.
  AVT03: AVT03 (denosumab) is a recombinant fully human IgG2 monoclonal antibody to RANKL to be administered as a subcutaneous injection. Subjects in this arm will receive AVT03 60mg administered s.c. on Day 1 and at Month 6. At Month 12, subjects in the AVT03 arm will receive a third dose of AVT03 60 mg.
- Prolia: Denosumab: Prolia (denosumab) is a recombinant fully human IgG2 monoclonal antibody to RANKL developed to be administered as a subcutaneous injection.
  Subjects will receive 60mg of commercially available US-Prolia, administered s.c on Day 1 and Month 6. At Month 12, subjects in the Prolia treatment group will be re-randomized in a 1:1 ratio to receive either:
  * AVT03 60 mg administered s.c. on Day365.
  * Prolia 60 mg administered s.c. on Day365.
- Prolia/AVT03 (Month 12 to Month18): Participants re-randomized on Month 12 from Prolia to AVT03 arm
Period: Baseline to Month 12
Arm/Group | AVT03 | Prolia | Prolia/AVT03 (Month 12 to Month18)
Started | 266 | 266 | 0
Completed | 242 | 244 | 0
Not Completed | 24 | 22 | 0
Not completed — Adverse Event | 7 | 2 | 0
Not completed — Death | 3 | 1 | 0
Not completed — Withdrawal by Subject | 11 | 16 | 0
Not completed — Protocol Violation | 2 | 3 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Month 12 to Month 18
Arm/Group | AVT03 | Prolia | Prolia/AVT03 (Month 12 to Month18)
Started | 242 (Participants randomized on baseline to AVT03 and kept on this arm after Month 12.) | 122 (Participants from Prolia arm re-randomized on Month 12 to Prolia Arm.) | 122 (Participants from Prolia arm re-randomized on Month 12 to AVT03 Arm)
Completed | 237 | 120 | 119
Not Completed | 5 | 2 | 3
Not completed — Death | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Other reasons | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- AVT03: AVT03 is a proposed biosimilar for Prolia.
  AVT03: AVT03 (denosumab) is a recombinant fully human IgG2 monoclonal antibody to RANKL to be administered as a subcutaneous injection. Subjects in this arm received AVT03 60mg administered s.c. on Day 1 and at Month 6. At Month 12, subjects in the AVT03 arm received a third dose of AVT03 60 mg.
- Prolia: Denosumab: Prolia (denosumab) is a recombinant fully human IgG2 monoclonal antibody to RANKL developed to be administered as a subcutaneous injection.
  Subjects will receive 60mg of commercially available US-Prolia, administered s.c on Day 1 and at Month 6. At Month 12, subjects in the Prolia treatment group will be re-randomized in a 1:1 ratio to receive either:
  * AVT03 60 mg administered s.c. on Day365.
  * Prolia 60 mg administered s.c. on Day365.
- Total: Total of all reporting groups
Arm/Group | AVT03 | Prolia | Total
Number analyzed (Participants) | 266 | 266 | 532
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (6.94) | 64.5 (7.04) | 64.9 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 266 | 266 | 532
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 11 | 24
  White | 246 | 249 | 495
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 5 | 6 | 11
Region of Enrollment [Number; unit: participants]
  Czechia | 28 | 33 | 61
  Poland | 144 | 144 | 288
  South Africa | 47 | 41 | 88
  Georgia | 33 | 37 | 70
  Bulgaria | 14 | 11 | 25
BMI at screening [Mean (Standard Deviation); unit: kg/m^2] | 25.12 (3.547) | 25.2 (3.605) | 25.16 (3.573)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in LS BMD at Month 12 to Demonstrate Comparable Efficacy of AVT03 and Prolia®.
Description: Percent Change From Baseline in LS BMD at Month 12 to demonstrate comparable efficacy of AVT03 and Prolia®.
Time Frame: Baseline to Month 12
Population: The number of evaluable subjects with data at Month 12 per group.
Measure: Least Squares Mean (Standard Error); unit: Percent Change From Baseline in LS BMD
Groups:
- Prolia: Denosumab: Prolia (denosumab) is a recombinant fully human IgG2 monoclonal antibody to RANKL developed to be administered as a subcutaneous injection.
  Subjects received 60mg of commercially available US-Prolia, administered s.c. on Day 1 and at Month 6. At Month 12, subjects in the Prolia treatment group were re-randomized in a 1:1 ratio to receive either:
  * Group 2a: Subjects will receive AVT03 60 mg administered s.c. on Day365.
  * Group 2b: Subjects will receive Prolia 60 mg administered s.c. on Day365.
Arm/Group | AVT03 | Prolia
Number analyzed (Participants) | 239 | 237
Percent Change From Baseline in LS BMD | 5.3 (0.870) | 5.18 (0.872)

2. Primary Outcome: To Demonstrate Comparable Profile of AVT03 and Prolia in Terms of Area Under the Percent Change From Baseline in Serum C-telopeptide of Type 1 Collagen (AUEC of %Cfb sCTX-1)
Time Frame: Baseline to Month 6
Population: The number of evaluable subjects with data at Month 12 per group.
Measure: Geometric Least Squares Mean (Standard Error); unit: percentage change from baseline*days
Groups:
- Prolia: Denosumab: Prolia (denosumab) is a recombinant fully human IgG2 monoclonal antibody to RANKL developed to be administered as a subcutaneous injection.
  Subjects received 60mg of commercially available US-Prolia, administered s.c on Day 1 and at Month 6. At Month 12, subjects in the Prolia treatment group were re-randomized in a 1:1 ratio to receive either:
  * AVT03 60 mg administered s.c. on Day365.
  * Prolia 60 mg administered s.c. on Day365.
Arm/Group | AVT03 | Prolia
Number analyzed (Participants) | 243 | 248
percentage change from baseline*days | 2345.55 (1.011) | 2342.87 (1.011)

3. Secondary Outcome: Percent Change From Baseline in LS BMD
Description: Percent change from Baseline in LS BMD at 6 and 18 months
Time Frame: Month 6, Month18
Reporting Status: Not Posted

4. Secondary Outcome: Percent Change From Baseline in Hip and Femoral Neck BMD
Description: Percent change from Baseline in hip and femoral neck BMD at Month 6, 12 and 18 months
Time Frame: Month 6, Month 12, Month 18
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of New Morphometric Vertebral Fractures
Description: Incidence of new morphometric vertebral fractures at 12 and 18 months
Time Frame: Month 12 and 18
Reporting Status: Not Posted

6. Secondary Outcome: Percent Change From Baseline in sCTX-1
Description: Percent change from Baseline in sCTX-1 at 3, 6, 9, 12 and 18 months
Time Frame: Month 3, Month 6, Month 9, Month 12 and Month 18
Reporting Status: Not Posted

7. Secondary Outcome: Incidence, Nature and Severity of Adverse Events Including Adverse Drug Reactions
Time Frame: Month 18
Reporting Status: Not Posted

8. Secondary Outcome: Frequency and Severity of Injection Site Reactions
Time Frame: Month 12
Reporting Status: Not Posted

9. Secondary Outcome: Frequency and Severity of Findings in Routine Safety Parameters
Time Frame: Month 18
Reporting Status: Not Posted

10. Secondary Outcome: Frequency and Titer of Anti-drug Antibodies and Frequency of Neutralizing Antibodies Against AVT03 and Prolia
Time Frame: Month 18
Reporting Status: Not Posted

11. Secondary Outcome: Serum Trough Concentration of AVT03 and Prolia
Time Frame: Month 18
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From baseline to Month 18
Groups:
- AVT03 (Baseline to Month 12): Randomized on Baseline to AVT03
- Prolia (Baseline to Month 12): Randomized on Baseline to Prolia
- AVT03 (Month 12 to Month18): Continuation on AVT03.
- Prolia/AVT03 (Month 12 to Month18): Re-randomized on Month 12 to AVT03
- Prolia/Prolia (Month 12 to Month18): Re-randomized on Month 12 to Prolia
Arm/Group | AVT03 (Baseline to Month 12) | Prolia (Baseline to Month 12) | AVT03 (Month 12 to Month18) | Prolia/AVT03 (Month 12 to Month18) | Prolia/Prolia (Month 12 to Month18)
All-Cause Mortality (participants affected / at risk) | 3/266 | 1/266 | 1/242 | 0/122 | 0/122
Serious Adverse Events (participants affected / at risk) | 9/266 | 10/266 | 6/242 | 3/122 | 2/122
Other Adverse Events (participants affected / at risk) | 178/266 | 178/266 | 99/242 | 39/122 | 39/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVT03 (Baseline to Month 12) (N=266) | Prolia (Baseline to Month 12) (N=266) | AVT03 (Month 12 to Month18) (N=242) | Prolia/AVT03 (Month 12 to Month18) (N=122) | Prolia/Prolia (Month 12 to Month18) (N=122)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroidism primary (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erosive duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Infective myositis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVT03 (Baseline to Month 12) (N=266) | Prolia (Baseline to Month 12) (N=266) | AVT03 (Month 12 to Month18) (N=242) | Prolia/AVT03 (Month 12 to Month18) (N=122) | Prolia/Prolia (Month 12 to Month18) (N=122)
Abnormal clotting factor (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 7 (8) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Macrocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart failure with preserved ejection fraction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Factor XII deficiency (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye haematoma (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudophakia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cascade stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 8 (8) | 1 (1) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 6 (11) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Gastric mucosa erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Intestinal barrier dysfunction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Noninfective gingivitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 10 (10) | 8 (10) | 1 (1) | 1 (1) | 1 (2)
Malaise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic calcification (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic dysfunction-associated liver disease (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 9 (9) | 3 (3) | 2 (3) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 7 (7) | 4 (4) | 2 (2) | 2 (2) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 7 (7) | 2 (3) | 3 (3) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes virus infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 8 (9) | 11 (12) | 0 (0) | 1 (1) | 0 (0)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (4) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 23 (25) | 20 (23) | 9 (9) | 3 (3) | 2 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Oral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 4 (4) | 5 (5) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 32 (37) | 36 (44) | 7 (8) | 1 (1) | 8 (8)
Urinary tract infection (Infections and infestations) | 14 (16) | 5 (6) | 3 (3) | 3 (3) | 3 (3)
Viral infection (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Arthropod sting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3) | 6 (6) | 1 (1) | 2 (3)
Tooth fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 13 (13) | 15 (16) | 8 (8) | 3 (4) | 6 (6)
Adjusted calcium decreased (Investigations) | 14 (15) | 6 (6) | 8 (8) | 4 (4) | 0 (0)
Adjusted calcium increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Calcium ionised decreased (Investigations) | 7 (8) | 7 (8) | 6 (6) | 3 (4) | 2 (2)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coagulation factor increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Creatinine renal clearance increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis B core antibody positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Red blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cells urine positive (Investigations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 28 (34) | 23 (28) | 5 (5) | 1 (1) | 3 (3)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired fasting glucose (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 (16) | 9 (11) | 3 (3) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9) | 5 (5) | 1 (2) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arachnoid cyst (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 10 (11) | 9 (9) | 2 (2) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Trigeminal neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis noninfective (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocyturia (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (3) | 3 (4) | 0 (0) | 1 (1) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract inflammation (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Telangiectasia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria chronic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 12 (13) | 8 (8) | 2 (2) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phlebitis superficial (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/91/NCT05395091/Prot_SAP_000.pdf